CLINICAL TRIAL: NCT04695093
Title: Investigating the Impact of London's Ultra Low Emission Zone on Children's Respiratory Health
Brief Title: Children's Health in London and Luton (CHILL)
Acronym: CHILL
Status: Active, not recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: King's College London (Other); University of Edinburgh (Other); University of Bedfordshire (Other); University of Cambridge (Other); University of Southern California (Other)
Responsible Party: Sponsor
Other Study IDs: 239719
Record Dates: First submitted 2020-10-26; First posted 2021-01-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Pollution; Exposure; Respiratory Disease; Child Development
Keywords: respiratory disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal/saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- London (intervention): 1606 children aged 6-9 yrs old, recruited in 44 London primary schools (years 2-4) within the Central London ULEZ area
  Interventions: Other: Ultra Low Emission Zone (ULEZ)
- Luton (comparison): 1706 children aged 6-9 yrs old, recruited in 41 Luton and Dunstable primary schools (years 2-4)

INTERVENTIONS:
Other: Ultra Low Emission Zone (ULEZ) — The ULEZ comprises a Central London zone, implemented on 8th April 2019, within which polluting vehicles are subject to a charge. Using number plate recognition technology, a daily penalty charge notice is issued for vehicles entering this central zone not meeting the standard of Euro 4 for petrol, Euro 6/VI for diesel, and Euro for motorcycles.
  The ULEZ will subsequently be extended to include:
  1. In 2020, a London-wide ULEZ for heavy duty vehicles (HDV) within the LEZ boundary (green zone). HDVs not meeting Euro 6 standard will be charged daily.
  2. In 2021, an Inner London ULEZ area for all light duty vehicles (LDV) within the boundary of the North and South Circular Roads (yellow zone). Vehicles not meeting the above criteria will be charged daily as for the Central London area.
  Other Names: Clean Air Zone
  Groups: London (intervention)

SUMMARY:
Investigating the impact of London's Ultra Low Emission Zone on children's respiratory health

DETAILED DESCRIPTION:
Strong evidence links urban air pollution to restrictions in children's lung growth and development and other adverse effects, including increases in respiratory and allergy symptoms, respiratory infections, asthma, and health care use. Effective interventions are urgently needed that reduce air pollution and improve child health. Low Emission Zones (LEZ) are becoming widespread but are expensive to implement and of unproven health benefit. London has some of the worst air pollution in Europe. London's Ultra Low Emission Zone (ULEZ) is the central component of London's air quality strategy. Its implementation provides a unique opportunity to test the impact of a city-wide LEZ on children's health.

The intervention:

The ULEZ is an area within which all vehicles must meet exhaust emission standards or pay a daily charge to travel. It will be implemented and paid for by Transport for London. Starting in 2019, the ULEZ will initially cover London's central Congestion Charging Zone, an area bounded by the London Inner Ring Road, that includes the City of London plus adjacent areas of eight radially adjoining Boroughs. It is projected to deliver for central London by 2020 emission reductions of -49% for NOx; - 47% for NO2; and -11% for PM10. Subject to consultation, the ULEZ will subsequently extend to include an inner London area (within London's North and South Circular roads), and a London-wide area, for heavy vehicles only.

Questions:

1. What is the impact of the ULEZ on children's lung growth (the primary outcome)?
2. What is the impact of the ULEZ on secondary outcomes, including self-reported symptoms, respiratory infection, health care use and costs?
3. Does the ULEZ reduce health inequalities? 4) Is the ULEZ good value for money?

Study design:

Quasi-experimental study using a parallel cohort design. Population: 1520 children aged 6-9 yrs old, recruited in 26 London primary schools (school years 2, 3 and 4) in London's Central Ultra Low Emission Zone. Intervention: Ultra Low Emission Zone Comparison: 1520 children aged 6-9 yrs old, recruited in 26 primary schools (school years 2, 3 and 4) in Luton, matched for ethnicity, deprivation and baseline air quality.

Outcome: PRIMARY: Lung function growth (post-bronchodilator forced expiratory volume in one second (FEV1) measured by high quality spirometry at sequential annual school visits over four years. SECONDARY: Forced vital capacity (FVC), exhaled nitric oxide (FeNO), quality of life, respiratory infections, health care use, health costs.

Sample size:

To detect a 15ml/year FEV1 difference between central and outer London cohorts at 90% power and 0.05 significance requires children in each cohort, inflated to allow for clustering effect of schools, spirometry success, child and school attrition, and pre-specified sub group analyses, giving a total of 3120 children (60 children from 26 schools in each cohort).

Duration: 6 years Air quality data: Modeled exposures by London Air Quality Network Data management: NIHR accredited Pragmatic Clinical Trials Unit Analysis: Interaction analysis controlling for effect modifiers (eg passive smoke; ethnicity); health economic cost consequence analysis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for schools:

  * Primary schools within, or with catchment areas that include, the Central London ULEZ.
  * Primary schools within the Borough of Luton and town of Dunstable.
  * State or independent sectors.

Inclusion criteria for children:

• Children attending a study school, in years 2, 3, or 4, at study inception.

Exclusion Criteria:

* Exclusion criteria for schools:

  * Schools that are not primary schools within the above boundaries.

Exclusion criteria for children:

* Children with learning or physical disabilities sufficient for them to be unable to give informed assent to the study, or to carry out study procedures.
* Children with major lung disease (not including asthma).

Ages: 9 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 6-9 yrs old, recruited in 40 London primary schools (years 2, 3, 4) within the Central London ULEZ area
  and
  Children aged 6-9 yrs old, recruited in 40 Luton primary schools (years 2, 3 4).
Sampling Method: Non-Probability Sample
Enrollment: 3312 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Lung function growth as change in forced expiratory volume in one second (FEV1) per year | Four years, 2018 -2021
  Measured by annual spirometry, as annual change in FEV1/year over 4 years

SECONDARY OUTCOMES:
Air quality, nitrogen dioxide (NO2) concentration derived from the the KCLUrban dispersion model | Four years, 2018 -2021
  Annual nitrogen dioxide (NO2) concentration (micrograms/cubic meter NO2)
Air quality, oxides of nitrogen (NOx) concentration derived from the KCLUrban dispersion model | Four years, 2018 -2021
  Annual oxides of nitrogen (NOx) concentration (micrograms/cubic meter NOx)
Air quality, particulate matter diameter <2.5microns derived from the KCLUrban dispersion model | Four years, 2018 -2021
  Annual particulate matter diameter <2.5microns (PM2.5) concentration (micrograms/cubic meter PM2.5)
Air quality, particulate matter diameter <2.5microns derived from the KCLUrban dispersion model | Four years, 2018 -2021
  Annual particulate matter diameter <2.5microns (PM2.5) concentration (micrograms/cubic meter PM10)
Lung capacity as FVC (forced vital capacity) | Four years, 2018 -2021
  Measured by annual spirometry, as FVC in litres
Annual prevalence of wheeze, as proportion (%) of respondents reporting wheeze | Four years, 2018 -2021
  International Study of Asthma and Allergies in Childhood (ISAAC) questionnaire for 6-7 year olds
Annual prevalence of eczema, as proportion (%) of respondents reporting eczema | Four years, 2018 -2021
  International Study of Asthma and Allergies in Childhood (ISAAC) questionnaire for 6-7 year olds
Annual prevalence of rhinitis, as proportion (%) of respondents reporting rhinitis | Four years, 2018 -2021
  International Study of Asthma and Allergies in Childhood (ISAAC) questionnaire for 6-7 year olds
Annual prevalence/participant of upper respiratory tract infections | Four years, 2018 -2021
  Electronic download of coded NHS health record data
Annual prevalence/participant of lower respiratory tract infections | Four years, 2018 -2021
  Electronic download of coded NHS health record data
Physical activity, as Percentage time in Moderate to Vigorous Physical activity per participant (MVPA) | Four years, 2018 -2021
  Annual hip accelerometer records of participants, measured over one week
Annual health care use per participant | Four years, 2018 -2021
  Electronic download of coded NHS health record data
Annual health care costs per participant | Four years, 2018 -2021
  Electronic download of coded NHS health record data and self report data
Cognitive function as average Movement Time in seconds (MT) on the Clinical Kinematic Assessment Test | Three years, 2019 -2021
  Annual Clinical Kinematic Assessment Test
Child Quality of Life as score out of 40 | Four years, 2018 -2021
  Annual parental completion of the CHU9D (Child Health Utility 9 Dimension) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mays Jawad, PhD, Study Director — Queen Mary University of London
Locations (1):
- Queen Mary University of London, London, United Kingdom

REFERENCES:
- [Derived] Tsocheva I, Scales J, Dove R, Chavda J, Kalsi H, Wood HE, Colligan G, Cross L, Newby C, Hall A, Keating M, Sartori L, Moon J, Thomson A, Tomini F, Murray A, Hamad W, Tijm S, Hirst A, Vincent BP, Kotala P, Balkwill F, Mihaylova B, Grigg J, Quint JK, Fletcher M, Mon-Williams M, Wright J, van Sluijs E, Beevers S, Randhawa G, Eldridge S, Sheikh A, Gauderman W, Kelly F, Mudway IS, Griffiths CJ. Investigating the impact of London's ultra low emission zone on children's health: children's health in London and Luton (CHILL) protocol for a prospective parallel cohort study. BMC Pediatr. 2023 Nov 4;23(1):556. doi: 10.1186/s12887-023-04384-5. PMID 37925402